CLINICAL TRIAL: NCT06908460
Title: The Link Between the Training of Nursing Home Professionals and the Quality of Life of Residents With Parkinson's Disease
Brief Title: Training of Nursing Home Professionals and Quality of Life of Residents With Parkinson's Disease
Acronym: PARK-EHPAD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: France Parkinson Association (Other)
Responsible Party: Principal Investigator, Céline PISCICELLI, PhD, The Link Between the Training of Nursing Home Professionals and the Quality of Life of Residents With Parkinson's Disease., University Hospital, Grenoble
Other Study IDs: PARK-EHPAD; 2024-A02733-44 (Other: ID RCB)
Record Dates: First submitted 2025-03-13; First posted 2025-04-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; nursing home; training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The complexity of medication treatments and the diversity of symptoms in Parkinson's disease (PD) require healthcare professionals to have specific knowledge of the disease in order to manage symptoms optimally and on an individualized basis. This becomes even more important as the disease progresses due to the evolution of symptoms into fluctuating motor and non-motor manifestations. People with PD residing in nursing homes (EHPADs) often have multiple comorbidities, making care even more complex. A lack of specific knowledge among healthcare professionals in EHPADs can expose residents to an increased risk of complications and dependence, affecting their quality of life. Additionally, the complex symptoms of these residents can create concerns for care teams, which can act as a barrier to admitting this population of elderly people into these institutions. Thus, training professionals who care for and support elderly individuals with PD is a priority to optimize the healthcare journey for people with Parkinson's.

Interventions aimed at improving care quality are often implemented without evaluating their impact or using methodologies that do not provide scientific evidence justifying their generalization. Evaluating these interventions is essential to develop effective interventions within the healthcare system, contributing both to the improvement of care quality and to health policy. These interventions should undergo an evaluation of their positive and negative effects before being generalized.

The PARK-EHPAD study aims to assess the link between the training of healthcare professionals and the quality of life of elderly individuals with PD living in EHPADs. Since 2015, the Parkinson's Expert Center (CEP) at CHU Grenoble-Alpes, in partnership with the Regional Health Agency (ARS), has provided specific training on the multidisciplinary management of PD for healthcare professionals in EHPADs in five departments of the Auvergne Rhône-Alpes (AURA) region-Isère, Savoie, Haute-Savoie, Drôme, and Ardèche. The hypothesis is that this theoretical training program improves staff knowledge on PD-related topics, which should lead to optimized practices and a clinically significant improvement in the quality of life (primary outcome) for people with PD residing in EHPADs.

The impact of training on professionals' knowledge will be assessed in a prior study (PARK-EHPAD PRO), an RNIPH-type study that began in October 2024. PARK-EHPAD PRO will evaluate the impact of training on knowledge, competence, and comfort in working with people with Parkinson's among healthcare professionals in EHPADs receiving the training. This study will strengthen the results of the observational PARK-EHPAD study, which focuses on the relationship between healthcare professionals' training and the quality of life of PD residents.

Among various secondary hypotheses, it is also predicted that this theoretical training program will improve not only knowledge but also the sense of competence (secondary outcome) of healthcare professionals, which should lead to an improvement in the quality of life at work (QVT) for these residents (secondary outcomes).

The results of the PARK-EHPAD study could have significant clinical implications for both the care pathway of people with PD and public health policy. For people with PD, better training for healthcare professionals in EHPADs, leading to optimized care practices, will improve comfort and the management of disability at advanced stages of the disease. This benefit could extend to residents, caregivers, and their wider circle.

Demonstrating a link between professional training and residents' quality of life in EHPADs would provide a strong argument for advocating the nationwide expansion of specific training programs to other CEPs. This would help optimize the healthcare journey for elderly individuals with PD (disability management) and improve the quality of life for healthcare professionals in EHPADs. Indeed, improving professionals' sense of competence, better disability management for residents, and improved satisfaction for residents and their families should lead to better quality of life at work for EHPAD staff. This perspective is essential in light of societal public health challenges related to the recruitment and retention of healthcare professionals in such institutions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Have a confirmed diagnosis of Parkinson's disease
* Reside in a nursing home (EHPAD) in the departments of 38, 73, 74, 26, and 07 in the AURA region
* Be able to cooperate and answer the questionnaires

Exclusion Criteria:

* Resident's opposition
* Subject to the provisions of articles L1121-5 to L1121-8 of the Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nursing home residents with Parkinson's disease
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-08-26 (Estimated); Study Completion 2027-08-26 (Estimated)

PRIMARY OUTCOMES:
Quality of Life-Alzheimer's Disease Scale (QOL-AD) | single visit, 1 hour
  The QOL-AD is a validated questionnaire assessing quality of life in patients with Alzheimer's disease. The scale ranges from 13 to 52, with higher scores indicating better quality of life.of life of residents with Parkinson's disease.

SECONDARY OUTCOMES:
Maslach Burnout Inventory (MBI) of healthcare professionals | single visit, 1 hour
  The MBI is a validated questionnaire assessing burnout in healthcare professionals. It consists of three subscales: Emotional Exhaustion (score range 0-54), Depersonalization (score range 0-30), and Personal Accomplishment (score range 0-48). Higher scores on Emotional Exhaustion and Depersonalization indicate higher burnout levels (worse outcome), whereas higher scores on Personal Accomplishment indicate lower burnout (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided